CLINICAL TRIAL: NCT05139576
Title: Practices of Vitamin D Supplementation Leading to Vitamin D Toxicity: Experience From a Tertiary Care Center of a Low Middle Income Country
Brief Title: Practices of Vitamin D Supplementation Leading to Vitamin D Toxicity
Status: Completed | Type: Observational
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Siraj Muneer, Resident, Aga Khan University Hospital, Pakistan
Other Study IDs: 2019-1973-5495
Record Dates: First submitted 2021-11-30; First posted 2021-12-01 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Vitamin D Toxicity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric Subjects and adults: Subjects were categorized into two age groups: <18 years (pediatric) and ≥18 years (adult).
  Interventions: Diagnostic Test: serum 25OHD testing
- Pediatrics and adults: Subjects were categorized into two age groups: <18 years (pediatric) and ≥18 years (adult).
  Interventions: Diagnostic Test: serum 25OHD testing

INTERVENTIONS:
Diagnostic Test: serum 25OHD testing — Subjects tested for serum 25OHD between April 2020 to March 2021 was reviewed daily and those with 25OHD levels >150 ng/ml were contacted via telephone.

SUMMARY:
To determine the frequency toxicity (>150 ng/ml) in subjects for 25-hydroxyvitamin D (25OHD) and evaluate the vitamin D (VD) supplements used by these subjects.

DETAILED DESCRIPTION:
This prospective cross-sectional study was conducted at the Section of Chemical Pathology, Department of Pathology and Laboratory Medicine, AKUH Karachi Pakistan after approval from Aga Khan University Hospital's Ethics Review Committee (ERC ID: 2019-1973-6924). Data of subjects tested for serum 25OHD between April 2020 to March 2021 was reviewed daily and those with 25OHD levels >150 ng/ml were contacted via telephone. Only the initial results of the subjects tested at Clinical Laboratory were included. Those with incomplete clinical history, 25OHD levels <150ng/ml, whose contact numbers were unavailable or not answering telephone calls were excluded. To maintain confidentiality all identifiers were removed, and study identity numbers were generated.

After explaining the reason for phone call, verbal informed consent was taken and clinical information of calcium and VD supplementation including prescribed or self-medicated, indications for prescription, formulation strength, total dosage, frequency, duration, and calcium status was collected on a structured clinical history forms. The hypercalcemia was labeled when serum calcium was >10.2 mg/dl.

Data analysis:

The statistical analysis was performed using the Microsoft Excel 2016. Subjects were categorized into two age groups: <18 years (pediatric) and ≥18 years (adult). Total doses of VD supplements were added to calculate cumulative supplementation and daily supplementation was calculated by dividing cumulative dose by duration of supplementation.

Descriptive statistics median (interquartile range, IQR) were calculated for numerical data while frequency (percentage) for categorical data. Frequencies of subjects with VD toxicity were derived and their correlates were evaluated in the both the age groups. Demographics (age and gender), calcium status of subjects, indications, formulation strengths, frequency, duration, cumulative and daily dose of supplementation were generated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects WITH serum 25OHD levels >150 ng/ml.
* Only the initial results.

Exclusion Criteria:

* Serum 25OHD levels <150ng/ml,
* Incomplete clinical history
* Whose contact numbers were unavailable
* Who were not answering telephone calls

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects tested for serum 25OHD
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Potential vitamin D toxicity | April 2020 to March 2021
  Frequency of potential vitamin D Toxicity and use of VD supplementation including prescribed or self-medicated, indications for prescription, formulation strength, total dosage, frequency and duration will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- The Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
To maintain confidentiality all identifiers were removed, and study identity numbers were generated. Individual data will not be shared

DOCUMENTS (3):
  • Study Protocol (2019-11-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT05139576/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT05139576/SAP_001.pdf
  • Informed Consent Form (2019-11-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT05139576/ICF_002.pdf